CLINICAL TRIAL: NCT02759926
Title: The Role of Bitter Taste Receptors Expressed in the Gastrointestinal Tract in Altering Food Intake and Gastrointestinal Motility
Brief Title: The Effect of Bitter Taste Receptor Agonists on The Gastrointestinal Tract, Hunger and Food Intake
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: BitterMotilityHungerFoodIntake
Record Dates: First submitted 2016-04-25; First posted 2016-05-03 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-04

CONDITIONS: Healthy; Obesity
Keywords: Healthy volunteers; Obesity; Bitter
MeSH Terms: conditions — Obesity | interventions — denatonium; Quinine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- Denatonium benzoate intragastric (Active Comparator): 1 µmol/kg bodyweight (10mM) was administered as a bolus into the stomach through a nasogastric feeding tube.
  Interventions: Drug: Denatonium benzoate
- Quinine hydrochloride intragastric (Active Comparator): 10 µmol/kg bodyweight (100mM) was administered as a bolus into the stomach through a nasogastric feeding tube.
  Interventions: Drug: Quinine hydrochloride
- Tap water intragastric (Placebo Comparator): An equal amount of tap water was administered as a bolus into the stomach through a nasogastric feeding tube.
  Interventions: Drug: Tap water
- Denatonium benzoate intraduodenal (Active Comparator): 1 µmol/kg bodyweight (10mM) was administered as a bolus into the proximal part of the duodenum through a nasogastric feeding tube.
  Interventions: Drug: Denatonium benzoate
- Quinine hydrochloride intraduodenal (Active Comparator): 10 µmol/kg bodyweight (100mM) was administered as a bolus into the proximal part of the duodenum through a nasogastric feeding tube.
  Interventions: Drug: Quinine hydrochloride
- Tap water intraduodenal (Placebo Comparator): An equal amount of tap water was administered as a bolus into the proximal part of the duodenum through a nasogastric feeding tube.
  Interventions: Drug: Tap water

INTERVENTIONS:
Drug: Denatonium benzoate
  Arms: Denatonium benzoate intraduodenal; Denatonium benzoate intragastric
Drug: Quinine hydrochloride
  Arms: Quinine hydrochloride intraduodenal; Quinine hydrochloride intragastric
Drug: Tap water
  Arms: Tap water intraduodenal; Tap water intragastric

SUMMARY:
In this study, the investigators aimed at evaluating the role of bitter taste receptors in the gastrointestinal tract (GIT). Intragastric or intraduodenal administration of denatonium benzoate (DB) or quinine hydrochloride were compared with placebo administration for their effects on lingual sensitivity, gastrointestinal motility (both in the fasted and fed state), gut hormone release (motilin, ghrelin, glucagon-like peptide-1 (GLP-1) and cholecystokinin (CCK)) and food intake. Differences between lean and obese subjects will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* BMI>30 kg/m² for the obese volunteers
* BMI<30 kg/m² for the lean volunteers
* Subject is capable and willing to give informed consent
* Female volunteers of child bearing potential must use oral, injected or implanted hormonal methods of contraception

Exclusion Criteria:

* Female volunteer is pregnant or breastfeeding
* Gastrointestinal diseases, major abdominal surgery
* Major psychiatric illnesses
* Volunteers that use drugs affecting the GIT or the central nervous system (CNS)
* Volunteers that suffer from diabetes mellitus
* Volunteers suffering from an endocrine disease such as diabetes, Cushing's disease, Addison's disease, hypothalamic tumor…
* Volunteers that have undergone surgical procedure for weight loss

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Estimated)
Dates: Start 2011-08; Primary Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in gastrointestinal motility measured by antroduodenal high-resolution manometry | 2 hours after administration, continuous measurement with high resolution manometry

SECONDARY OUTCOMES:
Change in gut hormone release measured by specific radioactive immunoassays | 2 hours after administration, blood sample every 10 min
Change in food intake measured by the caloric content of the meal | ad libitum food intake for 1 hour, 40 min after administration
Change in subjective hunger and satiety scores measured by visual analogue scales of 100 mm | 2 hours after administration, assessment every 5 min

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, Prof, Principal Investigator — Universitaire Ziekenhuizen KU Leuven

REFERENCES:
- [Derived] Deloose E, Janssen P, Corsetti M, Biesiekierski J, Masuy I, Rotondo A, Van Oudenhove L, Depoortere I, Tack J. Intragastric infusion of denatonium benzoate attenuates interdigestive gastric motility and hunger scores in healthy female volunteers. Am J Clin Nutr. 2017 Mar;105(3):580-588. doi: 10.3945/ajcn.116.138297. Epub 2017 Feb 1. PMID 28148502